CLINICAL TRIAL: NCT00085150
Title: Pediatric Phase I Trial of LMB-2 for Refractory CD25-Positive Leukemias and Lymphomas
Brief Title: LMB-2 Immunotoxin in Treating Young Patients With Relapsed or Refractory Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000367333; NCI-04-C-0168; NCI-5903; NCT00082004 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2007-02

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult T-cell leukemia/lymphoma; recurrent childhood acute lymphoblastic leukemia; childhood Burkitt lymphoma; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; relapsing chronic myelogenous leukemia; acute undifferentiated leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Recurrence; Leukemia, Biphenotypic, Acute | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin

INTERVENTIONS:
Biological: LMB-2 immunotoxin

SUMMARY:
RATIONALE: LMB-2 immunotoxin can locate cancer cells and kill them without harming normal cells.

PURPOSE: This phase I trial is studying the side effects and best dose of LMB-2 immunotoxin in treating young patients with relapsed or refractory leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of LMB-2 immunotoxin in pediatric patients with CD-25 positive relapsed or refractory leukemia or lymphoma.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug, including the terminal elimination serum half-life, area under the curve, volume of distribution, and relationship to disease burden, in these patients.

Secondary

* Evaluate the immonogenicity of this drug in these patients.
* Determine response in patients treated with this drug.
* Determine changes in lymphocyte subsets, immunoglobulin levels, serum cytokines, and soluble cytokine receptor levels in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive LMB-2 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression, neutralizing antibodies (i.e., > 75% of the activity of 1 µg/mL of LMB-2 immunotoxin), or unacceptable toxicity. Patients achieving complete remission (CR) receive 2 additional courses beyond CR. Patients with acute lymphoblastic leukemia also receive cytarabine and hydrocortisone intrathecally once monthly concurrent with restaging lumbar punctures.

Cohorts of 3-6 patients receive escalating doses of LMB-2 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, a total of 12 patients are treated at that dose level.

Patients are followed weekly for 1 month and then monthly thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Non-Hodgkin's lymphoma, including the following subtypes:

    * Lymphoblastic lymphoma
    * Burkitt's lymphoma
    * Large cell lymphoma
    * Adult T-cell leukemia/lymphoma
    * Cutaneous T-cell lymphoma
    * Peripheral T-cell lymphoma
  * Hodgkin's disease
  * Acute myeloid leukemia
  * Chronic myelogenous leukemia
  * Acute lymphoblastic leukemia (ALL)

    * More than 5% blasts in the bone marrow (i.e., M2 marrow classification)
  * Acute hybrid leukemia, including the following subtypes:

    * Mixed lineage leukemia
    * Biphenotypic leukemia
    * Undifferentiated leukemia
* CD25-positive (CD25+) disease, meeting 1 of the following criteria:

  * More than 15% of malignant cells are CD25+ by immunohistochemistry with anti-CD25 antibody
  * More than 30% of malignant cells from a site are CD25+ by fluorescence-activated cell sorting analysis
* Measurable or evaluable disease
* Relapsed or refractory disease after at least 1 standard chemotherapy regimen AND 1 salvage regimen
* No available alternative curative therapies
* Ineligible for or refused hematopoietic stem cell transplantation OR disease activity that prohibits the required time to identify a suitable stem cell donor
* No CNS leukemia or lymphoma, as evidenced by any of the following criteria:

  * Cerebrospinal fluid (CSF) WBC > 5/µl AND confirmation of CSF blasts
  * Cranial neuropathies secondary to underlying malignancy
  * CNS lymphoma detected by radiological imaging

    * Prior CNS involvement with no current evidence of CNS malignancy allowed
* No isolated testicular ALL

PATIENT CHARACTERISTICS:

Age

* 6 months to 21 years

Performance status

* ECOG 0-3 (≥ 12 years of age)
* Lansky 40-100% (< 12 years of age)

Life expectancy

* Not specified

Hematopoietic

* Pancytopenia due to disease allowed
* For patients without bone marrow involvement:

  * Absolute neutrophil count > 1,000/mm^3
  * Platelet count > 50,000/mm^3 (transfusion independent)

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 5 times upper limit of normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine clearance ≥ 60 mL/min OR
* Creatinine, meeting the following age-related criteria:

  * ≤ 0.8 mg/dL (≤ 5 years of age)
  * ≤ 1.0 mg/dL (6 to 10 years of age)
  * ≤ 1.2 mg/dL (11 to 15 years of age)
  * ≤ 1.5 mg/dL (> 15 years of age)
* Calcium 2.0-2.9 mmol/L

Cardiovascular

* Ejection fraction ≥ 45% by MUGA OR
* Shortening fraction ≥ 28% by echocardiogram

Pulmonary

* Oxygen saturation ≥ 90%

Other

* Sodium 130-150 mmol/L
* Potassium 3.0-5.5 mmol/L
* Magnesium 0.5-1.23 mmol/L
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant unrelated systemic illness that would preclude study participation
* No conditions that would preclude study compliance
* No serum that neutralizes > 75% of the activity of 1 μg/mL of LMB-2 immunotoxin in tissue culture (due to either anti-toxin or anti-mouse immunoglobulin G antibodies)
* No active graft-vs-host disease (i.e., off immunosuppression)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior autologous bone marrow transplantation (BMT) allowed
* At least 100 days since prior allogeneic BMT
* At least 1 week since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or epoetin alfa)

Chemotherapy

* At least 2 weeks since prior chemotherapy (4 weeks for nitrosoureas) except intrathecal chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed provided the dose has been stable for the past week and does not increase during study treatment

  * Tapering or discontinuation of steroids allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy unless < 10% of marrow is irradiated and measurable disease exists outside the radiation port

Surgery

* Not specified

Other

* Recovered from all prior therapy
* At least 30 days since prior investigational agents
* Concurrent oral supplementation to maintain normal electrolyte levels allowed
* No concurrent anticoagulation therapy for disease-related conditions
* No other concurrent investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Wayne, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - St. Jude Children's Research Hospital, Memphis, Tennessee